CLINICAL TRIAL: NCT05205187
Title: Multi-center and Multi-omics Mechanism Research of Gut Microbiota and Metabonomics in Borrmann Type IV Gastric Cancer
Brief Title: Gut Microbiota and Metabonomics
Acronym: MBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); The Second Hospital of Shandong University (Other); The General Hospital of Fushun Mining Bureau (Unknown); The fourth People's Hospital of Changzhou (Unknown); The First People's Hospital of Jingzhou (Other)
Responsible Party: Principal Investigator, Kai Li, Deputy Director of surgical Oncology, First Hospital of China Medical University
Other Study IDs: Metabonomics
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Stomach Neoplasms; Gut Microbiota; Metabolomics
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy group: Healthy people in the community.
  Interventions: Procedure: Healthy control specimen collection
- Non-Borrmann IV group: Patients with Borrmann types I, II and III gastric cancer.
  Interventions: Procedure: Non-Borrmann IV patient specimen collection
- Borrmann IV group: Patients with Borrmann type IV gastric cancer.
  Interventions: Procedure: Borrmann IV patient specimen collection

INTERVENTIONS:
Procedure: Healthy control specimen collection — Collecting blood and feces from healthy population.
  Groups: Healthy group
Procedure: Non-Borrmann IV patient specimen collection — Collecting blood, feces and gastric cancer tissues from Non-Borrmann IV patients.
  Groups: Non-Borrmann IV group
Procedure: Borrmann IV patient specimen collection — Collecting blood, feces and gastric cancer tissues from Borrmann IV patients.
  Groups: Borrmann IV group

SUMMARY:
To evaluate the correlation between gut microbiota and metabolites in Borrmann type IV gastric cancer; To find the effects of microflora and metabolites on target organs; To detect the mechanism of key flora and metabolite by in vitro and in vivo experiments; To construct models of gut microbiota and metabonomics by machine learning.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign informed consent.
2. Borrmann classification of gastric cancer is determined by more than 2 pathologists.
3. Patients with BMI 24-28.
4. Karnofsky (KPS) score >80.

Exclusion Criteria:

1. Patients who take any aspirin, antibiotics, prebiotics, or probiotics within 4 weeks and steroids or immunosuppressants within 6 months prior to specimen collection.
2. Patients who complicate with other malignant tumors.
3. Patients who complicate with diabetes, hypertension, heart disease and infectious diseases.
4. Patients who complicate with inflammatory bowel disease or irritable bowel syndrome.
5. Patients with metastasis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population will be selected from community samples. Non-Borrmann IV and Borrmann IV patients will be selected from Department of Oncology in hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants' characteristics | 1 day
  To obtain participants' characteristics, including age, gender, alcohol consumption, body mass index, smoking, medications.
Microbial community structure | 1 day
  To assess participants' microbiome composition in faecal samples, inclding microbial diversity and richness.
Metabolite composition | 1 day
  To measure the metabolite profiles in participants' faecal samples and serum samples, involving Bile acids, short chain fatty acids, TMAO and related metabolites, amino acids, fatty acids, organic acids, flavonoids, plant hormones, neurotransmitters.
Microbes-metabolites correlations | 1 day
  To assess the correlations of gut microbiota and metabolites by Spearman's correlation analysis.
Response of target organ | 1 day
  To find the effects of microflora and metabolites on target organ by transcriptome sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Li, MD, Principal Investigator — First Hospital of China Medical University
Locations (6):
- China (6):
  - The fourth People's Hospital of Changzhou, Changzhou, Jiangsu
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - The General Hospital of Fushun Mining Bureau, Fushun, Liaoning
  - First Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The Second Hospital of Shandong University, Ji'nan, Shandong